CLINICAL TRIAL: NCT01395953
Title: Double-blind Trial of Buspirone for the Treatment of Anxiety in Youth With Autism Spectrum Disorders
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was withdrawn due to competing research interests and slow recruitment.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Gagan Joshi, Assistant Professor of Psychiatry, Harvard University, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-P-000703
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: Buspirone; Buspar; Autism Spectrum Disorders; Pervasive Developmental Disorders; Children; Adolescents; Anxiety
MeSH Terms: conditions — Autism Spectrum Disorder; Child Development Disorders, Pervasive; Anxiety Disorders | interventions — Buspirone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buspirone (Active Comparator)
  Interventions: Drug: Buspirone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buspirone — Children with Autism Spectrum Disorders will receive buspirone or matched placebo. Buspirone will be titrated to the maximum daily dose during the first four weeks of the trial (dose titration phase). Week 4 onwards subjects will be maintained on maximum achieved dose till the end of the trial (dose maintenance phase). During the titration phase total dose of buspirone will be increased at each visit by 5mg and on the 4th day after each visit by 5mg.
  Other Names: Buspar
  Arms: Buspirone
Drug: Placebo — Children with Autism Spectrum Disorders will receive buspirone or matched placebo. Buspirone will be titrated to the maximum daily dose during the first four weeks of the trial (dose titration phase). Week 4 onwards subjects will be maintained on maximum achieved dose till the end of the trial (dose maintenance phase). During the titration phase total dose of buspirone will be increased at each visit by 5mg and on the 4th day after each visit by 5mg.
  Arms: Placebo

SUMMARY:
The main objective of this exploratory 8 week pilot study is to evaluate the safety and efficacy of buspirone for the treatment of anxiety in youth (ages 6-17 years) with autism spectrum disorders. The study results will be used to generate hypotheses for a larger randomized controlled clinical trial with explicit hypotheses and sufficient statistical power.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants between 6 and 17 years of age.
* Fulfills diagnosis of autism spectrum disorders by meeting DSM-IV-TR PDD diagnostic criteria of autistic disorder, Asperger's disorder, or PDD-NOS as established by clinical diagnostic interview.
* Participants with a score of ≥60 on the Anxiety/Depression subscale of Child Behavior Checklist (CBCL) and CGI-Anxiety severity of ≥4.
* Subjects can be on psychotropic drugs if they have been on the medication for at least 4 weeks prior to initiating study treatment and if they are on a stable dose.
* Subjects with disruptive behavior disorders, mood, or psychosis will be allowed to participate in the study provided they do not meet any exclusionary criteria.

Exclusion Criteria:

* Mental retardation (I.Q. <70)
* DSM-IV-TR PDD diagnosis of Rett's disorder, and childhood disintegrative disorder.
* History of active seizure disorder (EEG suggestive of seizure activity and/or history of seizure in last 1 month).
* Subjects with a medical condition or treatment that will either jeopardize subject safety or affect the scientific merit of the study, including: pregnant or nursing females, organic brain disorders, uncorrected hypothyroidism or hyperthyroidism, clinically significant abnormalities on ECG (e.g. QT prolongation, arrhythmia), history of renal or hepatic impairment.
* Clinically unstable psychiatric conditions or judged to be at serious suicidal risk.
* History of substance abuse (except nicotine of caffeine) within past 3 months or urine drug screen positive for substances of abuse.
* Any other concomitant medication with primary central nervous system activity other than stable regimens for >2 weeks.
* A non-responder or history of intolerance to buspirone, after treatment at an adequate dose and duration as determined by the clinician.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Reduction in Pediatric Anxiety Rating Scale (PARS) Score | baseline to 8 weeks
  Primary outcome measure of efficacy will be assessed by reduction in anxiety symptom severity as measured by change from baseline. Responders are defined as ≥30% reduction in the Pediatric Anxiety Rating Scale (PARS).
Clinical Global Impression-Anxiety (CGI-Anxiety) Improvement Score | baseline to 8 weeks
  Primary outcome measure of efficacy will be assessed by reduction in anxiety symptom severity as measured by Clinical Global Impression-Anxiety (CGI-Anxiety). Responders are defined as a score of ≤2 on the improvement subscale (i.e., "much" or "very much improved").

CONTACTS AND LOCATIONS:
Overall Officials: Gagan Joshi, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States